CLINICAL TRIAL: NCT05850260
Title: Effect of Providing a Personal McGrath Video Laryngoscope to Anesthesiologists for All Intubations in the Operating Room: a Multicentre Prospective Observational, Before-after Study
Brief Title: McGrath Video Laryngoscope for All Intubations in the Operating Room
Acronym: VIDEO-SURG
Status: Completed | Type: Observational
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Associate Profesor, Hospital Clinico Universitario de Santiago
Other Study IDs: VIDEOLAR-SURGERY
Record Dates: First submitted 2023-04-18; First posted 2023-05-09 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-07

CONDITIONS: Intubation Complication
Keywords: diificult intubation; videolaryngoscope; airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Macintosh laryngoscope: During the pre-implementation period (6 months), the 35 assigned attending anesthetists will perform all tracheal intubations in the operation room according to the standard of care using the standard Macintosh direct laryngoscope as a first intubation option
  Interventions: Device: Macintosh laryngoscope
- McGrath Mac videolaryngoscope: During the post-implementation period (6 months), the 35 assigned attending anesthetists will perform all tracheal intubations using their personal McGrath Mac videolaryngoscope as a first intubation option
  Interventions: Device: Videolaryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscope — During the pre-implementation period (6 months), the 35 assigned attending anesthetists will perform all tracheal intubations in the operation room according to the standard of care using the standard Macintosh direct laryngoscope as a first intubation option
  Groups: Macintosh laryngoscope
Device: Videolaryngoscope — During the post-implementation period (6 months), the 35 assigned attending anesthetists will perform all tracheal intubations using their personal McGrath Mac videolaryngoscope as a first intubation option.
  Groups: McGrath Mac videolaryngoscope

SUMMARY:
Tracheal intubation is a very common procedure performed in the operating room. The usual intubation technique in the operating room is based on direct laryngoscopy, using a standard Macintosh laryngoscope. Although in most patients there are no complications during intubation, more than 90% of difficult tracheal intubations in the operate room are unpredictable, and several authors, recommend the universal use of the videolaryngoscope for all intubations, using as the first intubation option regardless of whether the patient has predictors of a difficult airway or no.The authors do not know whether providing a own videolaryngoscope to each anesthesiologist to use as the first option for intubation in all patients who need it in the operating room improves the percentage of patients with easy intubation and decrease the incidence of complications.

DETAILED DESCRIPTION:
Tracheal intubation is a very common procedure performed in the operating room. The usual intubation technique in the operating room is based on direct laryngoscopy, using a standard Macintosh laryngoscope. Although in most patients there are no complications during intubation, more than 90% of difficult tracheal intubations in the operate room are unpredictable, and several authors, recommend the universal use of the videolaryngoscope for all intubations, using as the first intubation option regardless of whether the patient has predictors of a difficult airway or no. The authors do not know whether providing a personal videolaryngoscope to each anesthesiologist to use as the first option for intubation in all patients who need it in the operating room improves the percentage of patients with easy intubation and decrease the incidence of complications.

The VIDEOLAR-SURGERY trial is a prospective, observational, open-label, multicenter study, with before-after analysis. Consecutive patients requiring tracheal intubation for an elective o urgent surgical intervention from a period of 14 months by one of the 35 researcher's anesthesiologists assigned will be recruited. In the pre-implementation period (6 months), the 35 anesthesiologists will perform all tracheal intubations using the standard Macintosh direct laryngoscope as a first intubation option. During the implementation period (2 months), a personal McGrath videolaryngoscope will be provided to each anesthesiologist to train in its use. During the post-implementation period (6 months), the 35 anesthesiologists will perform all tracheal intubations using their personal McGrath Mac videolaryngoscope as a first intubation option. The main objective is to evaluate whether the use of a own McGrath videolaryngoscope by anesthesiologists, as the first intubation option, improves the percentage of patients with easy intubation compared with the standard Macintosh laryngoscope. Secondary objectives are to compare incidence of first-attempt intubation, laryngoscopic vision, need of adjuvant airway devices, difficulty, and complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients who need to be tracheal intubated for a surgical intervention in the surgical area.

Exclusion Criteria:

* Patients who are intubated in a place other than the surgical area (Intensive Care, Emergency, Hospitalization floor) will not be included.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who need to be tracheal intubated for an elective o urgent surgical intervention from a period of 14 months by one of the 35 anesthesiologists assigned by the Anesthesiology Services of the 8 Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 5220 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
"easy intubation" | during intubation
  To compare "easy intubation" in the two study periods. "Easy intubation" defined as intubation at the first attempt, modified Cormack-Lehane grades of I or IIa and absence of need of adjuvant airway devices for intubation. (percentage)

SECONDARY OUTCOMES:
Intubations at the first attempt | during intubation
  To compare difference in the incidence of intubations at the first attempt in the two periods studied. (percentage)
Number of intubations attempts | during intubation
  To compare number of intubations attempts in the two periods studied
Modified Cormack-Lehane grade of glottic view | during intubation
  To compare Modified Cormack-Lehane grade of glottic view in the two periods studied Modified Cormack-Lehane grade of glottic view:I: full view of the glottis IIa: partial view of the glottis IIb: arytenoid or posterior part of the vocal cords just visible III: only epiglottis visible IV: neither glottis nor epiglottis visible
Need of adjuvant airway devices for intubation | during intubation
  To compare need of adjuvant airway devices for intubation in the two periods studied airway devices for intubation: bougie, videolaryngoscope, others)
Operator-assessed subjective difficulty | during intubation
  To compare degree of subjective difficulty experienced by the operator in the two periods studied.
  Subjective difficulty of intubation by means of a special analogue numerical scale from 0 to 10, where 0=no subjective difficulty and 10=maximal subjective difficulty
Complications during intubation | Participants will be followed from the beginning of the intervention to 30 minutes after the intervention
  To compare percentage of complications associated with the intubation in the two periods studied
Overall success rate intubation | During intubation
  To compare the difference overall success rate intubation (percentage) with the first device used in each period
Need to change the device for intubation | During intubation
  To compare the need to change the device for intubation in the two periods studied

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada Muñiz, M.D., Ph.D., Principal Investigator — University Clinical Hospital of Santiago de Compostela
Locations (1):
- Manuel Taboada, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data types: Deidentified participant data How to access data: Requests must be sent to manutabo@yahoo.es When available: With publication Additional Information Who can access the data: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose Mechanisms of data availability: With investigator support
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When available: With publication
Access Criteria: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose

REFERENCES:
- [Background] Hansel J, Rogers AM, Lewis SR, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adults undergoing tracheal intubation: a Cochrane systematic review and meta-analysis update. Br J Anaesth. 2022 Oct;129(4):612-623. doi: 10.1016/j.bja.2022.05.027. Epub 2022 Jul 9. PMID 35820934
- [Background] De Jong A, Sfara T, Pouzeratte Y, Pensier J, Rolle A, Chanques G, Jaber S. Videolaryngoscopy as a first-intention technique for tracheal intubation in unselected surgical patients: a before and after observational study. Br J Anaesth. 2022 Oct;129(4):624-634. doi: 10.1016/j.bja.2022.05.030. Epub 2022 Jul 8. PMID 35811139
- [Background] Cook TM, Boniface NJ, Seller C, Hughes J, Damen C, MacDonald L, Kelly FE. Universal videolaryngoscopy: a structured approach to conversion to videolaryngoscopy for all intubations in an anaesthetic and intensive care department. Br J Anaesth. 2018 Jan;120(1):173-180. doi: 10.1016/j.bja.2017.11.014. Epub 2017 Nov 21. PMID 29397126
- [Background] Cooper RM. Implementing universal videolaryngoscopy: how to do it and what to expect. Br J Anaesth. 2018 Jan;120(1):13-15. doi: 10.1016/j.bja.2017.11.017. Epub 2017 Nov 21. No abstract available. PMID 29397120
- [Derived] Taboada M, Estany-Gestal A, Rama-Maceiras P, Orallo MA, Bermudez M, Barreiro C, Gomez L, Amor M, Otero F, Fernandez J, Molins N, Amate JJ, Bascuas B, Rey R, Alonso MC, Castro MJ, Sarmiento A, Dos Santos L, Nieto C, Paredes S, Velasco A, Taboada C, Martin L, Campana D, Mosquera E, Novoa C, Varela S, da Silva L, Dominguez E, Bedoya A, Gomez AI, Estevez M, Martinez P, Sotojove R, Naveiro A, Diaz C, Ruido R, Miron P, Gonzalez M, Francisco C, Regueira J, Peiteado M, Eiras M, Paz E. Impact of universal use of the McGrath videolaryngoscope as the first option for all intubations in the operating room: The multicentre prospective before-after VIDEOLAR-SURGERY study protocol. Rev Esp Anestesiol Reanim (Engl Ed). 2025 Jan;72(1):101649. doi: 10.1016/j.redare.2024.101649. Epub 2024 Nov 12. PMID 39542091